CLINICAL TRIAL: NCT02612506
Title: A Randomized, Double-Blinded, Safety and Pharmacokinetic Study of Escalating Single Doses of Hepalatide in Healthy Volunteers
Brief Title: Safety and Pharmacokinetic Study of Hepalatide(L47) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai HEP Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: L47-Ia-01
Record Dates: First submitted 2015-09-16; First posted 2015-11-23 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2016-07

CONDITIONS: Hepatitis B， Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Drug and Narcotic Control

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Hepalatide (Experimental): Hepalatide 0.21mg, 0.525mg, 2.1mg, 4.2mg, 6.3mg, 8.4mg and 10.5mg
  Interventions: Drug: Hepalatide
- Placebo (Placebo Comparator): Placebo 0.525mg, 2.1mg, 4.2mg, 6.3mg, 8.4mg and 10.5mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hepalatide — There are seven cohorts as follows 0.21mg, 0.525mg, 2.1mg, 4.2mg, 6.3mg, 8.4mg and 10.5mg. Dose of 0.21mg is a pilot trial with no placebo. At each dose level, healthy volunteers will be received treatment drug by abdominal subcutaneous injection at the first day and monitored for 8 days.
  Other Names: treatment drug
  Arms: Hepalatide
Drug: Placebo — There are six cohorts as follows 0.525mg, 2.1mg, 4.2mg, 6.3mg, 8.4mg and 10.5mg. At each dose level, healthy volunteers will be received control drug by abdominal subcutaneous injection at the first day and monitored for 8 days.
  Other Names: control drug
  Arms: Placebo

SUMMARY:
To evaluate the safety and tolerability of Hepalatide(L47) and characterize the clinical pharmacokinetics in healthy volunteers.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, dose escalating, phase Ia trial, which will be conducted in No. 302 Hospital of China. There are seven cohorts at dose of 0.21mg, 0.525mg, 2.1mg, 4.2mg, 6.3mg, 8.4mg and 10.5mg. The first cohort with 0.21mg is an open test with no placebo as control. All other healthy volunteers will be randomized into Hepalatide or placebo group at 4:1 rate, and will be received drug by abdominal subcutaneous injection and will be observed for 8 days.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 45 years
* BMI Index between 19 and 25 (BMI=weight/height2)
* Normal previous history and physical exam
* No drug and alcohol abuse
* No illness in 4 weeks and no drug therapy in 2 weeks
* No blood donation or subject not sampled in 3 months
* Consistent and correct use of recommended methods of birth control for men and women
* Good compliance with study protocol
* Understand and agree to sign a consent form

Exclusion Criteria:

* Infection with HAV, HBV, HCV, HEV, HIV, EBV or CMV
* Abnormal and clinical significance test of physical examination, vital signs, blood routines, urine routines, liver and kidney functions, coagulation indicator, electrolyte, glucose, blood lipid, thyroid functions, chest X-Ray, ECG, B ultrasound of gallbladder, spleen and kidney, AFP ,and CEA
* Positive for anti-Pre-S1 antibody
* Women being pregnant or nursing, or with abnormal sex hormones, B ultrasound of ovaries/uterus proliferative diseases or breast mass
* Unable to quit smoking in trial
* Subject with little chance of enrollment (i.e. the weak)
* Subject not suitable to join the trial under other circumstances judged by investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Healthy participants with treatment-related adverse events as assessed by "guiding principle of grading standards for the adverse reactions in clinical trials of vaccine for prevention" or CTCAE v4.0 | half a year

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | half a year
Area under the plasma concentration versus time curve (AUC) | half a year
half-time | half a year
apparent volume of distribution | half a year

CONTACTS AND LOCATIONS:
Overall Officials: zhenman Wei, Principal Investigator — 302 Military Hospital
Locations (1):
- 302 Military Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No